CLINICAL TRIAL: NCT00881673
Title: A Single-Center, Randomized, Double-Masked, Placebo-Controlled Evaluation of the Efficacy of AL-38583 in the Reduction of Tear Eosinophil Count Following Conjunctival Allergen Challenge (CAC)
Brief Title: To Evaluate the Efficacy of AL-38583 in the Reduction of Tear Eosinophil Count Following Conjunctival Allergen Challenge
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-005
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Allergic Conjunctivitis
Keywords: Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic; Conjunctivitis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: AL38583 Ophthalmic Solution
- 2 (Active Comparator)
  Interventions: Drug: Maxidex
- 3 (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AL38583 Ophthalmic Solution — Topical ophthalmic
  Arms: 1
Drug: Maxidex — Topical ophthalmic
  Arms: 2
Drug: Vehicle — AL38583 Vehicle
  Arms: 3

SUMMARY:
The purpose of the study is to determine whether Al38583 Ophthalmic Solution is safe and effective in reducing tear eosinophil levels at 5-8 hours after Conjunctival Allergen Challenge (CAC).

ELIGIBILITY:
Inclusion Criteria:

* Have a positive bilateral CAC reaction (>2 itching and > conjunctival redness) to cat hair, cat dander, dust mites, cockroaches and/or dog dander within 10 minutes of instillation of the last titration of allergen at Visit 1

Exclusion Criteria:

* Have a known allergy to the study medication(s) or their components (ex., dexamethasone, benzalkonium chloride)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is mean change in tear eosinophil level at Visit 7 post-CAC from Visit 2 post-CAC. | 15 days

SECONDARY OUTCOMES:
Mean change in relative ratio of tear eosinophil and neutrophils at Visit 7 post-CAC from Visit 2 post-CAC | 15 days